CLINICAL TRIAL: NCT01247792
Title: A Time-series Intervention Analysis of End-of-life Decision-making in Patients With Sepsis-related Organ Failure
Brief Title: End-of-life Decision-making in Patients With Sepsis-related Organ Failure
Acronym: EIDECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Sepsis Control and Care, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Christiane Hartog, PD Dr med. Christiane Hartog, Center for Sepsis Control and Care, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EIDECS
Record Dates: First submitted 2010-11-11; First posted 2010-11-24 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Severe Sepsis
Keywords: sepsis; organ failure; end-of-life decisions; patient-centered communication
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Before" (No Intervention): No Intervention Observation of current practice
- "After" (Other): SOPs for decision-making and communication Assessment of practice after implementation of SOPs
  Interventions: Behavioral: SOPs for decision-making and communication

INTERVENTIONS:
Behavioral: SOPs for decision-making and communication — Development and implementation of SOPs for timely and interdisciplinary EOL-decisionmaking and a communication strategy with relatives which addresses participants, set-up, time-points, and content
  Arms: "After"

SUMMARY:
The care of patients with sepsis-related organ failure on the intensive care unit (ICU) often includes end-of-life decision (EOL-D) and communication of such decisions to relatives. This increases the psychological burden for caregiver and relatives.

The investigators intend to assess the prevalence and impact of EOL-D on ICU care-givers and relatives ("before") and to use this data to develop and implement standard operating procedures (SOPs) for improved decision-making and communication of these decisions ("after").

The hypothesis is that an improved communication strategy will reduce symptoms of burnout in caregivers and symptoms of anxiety and depression in relatives.

DETAILED DESCRIPTION:
BACKGROUND About half of patients with sepsis related organ failure die on the ICU, frequently after end-of-life decisions (EOL-D), i.e. the decision to withdraw or withhold life-supporting therapies or forgo cardiopulmonary resuscitation. Lack of SOPs about how to communicate and share EOL-decisionmaking among staff and to communicate EOL-D to relatives may increase burnout and anxiety in staff as well as relatives. Also, there is uncertainty about the role of patients' advance directives in EOL-Decision-making.

HYPOTHESES 1. SOPs for interdisciplinary EOL-decisions will alleviate staff burnout; 2. A structured strategy to communicate EOL-decisions to relatives will lead to reduced anxiety and depression in relatives 3 months after the event.

AIMS 1. to develop SOPs for EOL-decision-making which improve timeliness of EOL-D and involvement of interdisciplinary care-givers. 2. to develop a strategy how to communicate these EOL-D to relatives including a structured procedure for participants, set-up, times and content. These aims may be adapted according to the findings of the observation period.

CONDUCT The study is designed as an interrupted time series analysis ("before/after study") located on the mixed, neurological and medical ICUs of the Jena University Hospital. It is composed of 3 observation periods separated by phases of data analysis and implementation of changes in behavioral practice. After the first phase of observation and data analysis, SOPs including an improved communication strategy with relatives will be developed on the basis of the collected data. SOPs will be developed and implemented on participating ICUs. In the following second observation period data will be collected to assess changed procedures and primary endpoints. A third round of data analysis, interpretation and observation will enable to further adapt SOPs and achieve sustainability ("post-implementation phase").

ESTIMATED ENROLLMENT Enrollment of 180 staff members (physicians and nursing staff) and 90 relatives during each study phase

ELIGIBILITY:
Staff:

Inclusion Criteria:

* all physicians and nursing staff who treat patients with sepsis-related organ failure on participating ICUs who consent to participate

Exclusion Criteria:

* Decline to participate

Relatives:

* Relatives of patients with sepsis-related organ failure and EOL-D who consent to participate

Exclusion Criteria:

* Decline to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-08; Primary Completion 2014-09-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Symptoms of burnout by MBI score in ICU caregivers | once during observation period (1 year)
Symptoms of post-traumatic stress disorder by IES and HADS scores in relatives at 90 days | once during observation period (1 year)

SECONDARY OUTCOMES:
Psychological symptoms by IES, HADS or MBI subscales in caregivers or relatives, respectively | once during the observation period (1 year)
Characteristics of patients with and without end-of-life decisions (EOL-D) including time periods (time until EOL-D, time between EOL-D until death or discharge) and 28-day and 90-day mortality rates | until death or discharge from the ICU
Prevalence and characteristics of EOL-D | until death or discharge from the ICU
Prevalence and characteristics of patients' advance directives | until death or discharge from the ICU
characteristics of EOL-D communication with relatives | ICU stay
Prevalence of request for "Ethik Konsil" (counseling by an external ethical review board) | until death or discharge from the ICU
direct costs of treatment of survivors and non-survivors | until death or discharge from the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Christiane S Hartog, MD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Jena University Hospital
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany

REFERENCES:
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Background] Embriaco N, Papazian L, Kentish-Barnes N, Pochard F, Azoulay E. Burnout syndrome among critical care healthcare workers. Curr Opin Crit Care. 2007 Oct;13(5):482-8. doi: 10.1097/MCC.0b013e3282efd28a. PMID 17762223
- [Result] Schwarzkopf D, Westermann I, Skupin H, Riedemann NC, Reinhart K, Pfeifer R, Fritzenwanger M, Gunther A, Witte OW, Hartog CS. A novel questionnaire to measure staff perception of end-of-life decision making in the intensive care unit--development and psychometric testing. J Crit Care. 2015 Feb;30(1):187-95. doi: 10.1016/j.jcrc.2014.09.015. Epub 2014 Sep 20. PMID 25311265
- [Result] Hartog CS, Schwarzkopf D, Riedemann NC, Pfeifer R, Guenther A, Egerland K, Sprung CL, Hoyer H, Gensichen J, Reinhart K. End-of-life care in the intensive care unit: a patient-based questionnaire of intensive care unit staff perception and relatives' psychological response. Palliat Med. 2015 Apr;29(4):336-45. doi: 10.1177/0269216314560007. Epub 2015 Jan 29. PMID 25634628